CLINICAL TRIAL: NCT06233461
Title: A Phase 2b, Multicenter, Randomized, Double-Blind Induction, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of Oral TAK-279 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Study on the Safety of TAK-279 and Whether it Can Reduce Inflammation in the Bowel of Participants With Moderately to Severely Active Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-279-CD-2001; 2023-506704-14-00 (EU CTIS Number: Abbreviated EU CT Number); jRCT2051240050 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy; Latitude CD, Latitude Research Program
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TAK-279 Dose 1 (Experimental): Participants will be randomized to receive TAK-279 Dose 1 capsules with TAK-279 placebo-matching capsule orally.
  Interventions: Drug: TAK-279; Drug: Placebo
- TAK-279 Dose 2 (Experimental): Participants will be randomized to receive TAK-279 Dose 2 capsules with TAK-279 placebo-matching capsule orally.
  Interventions: Drug: TAK-279; Drug: Placebo
- TAK-279 Dose 3 (Experimental): Participants will be randomized to receive TAK-279 Dose 3 capsules orally.
  Interventions: Drug: TAK-279
- Placebo (Experimental): Participants will be randomized to receive TAK-279 placebo-matching capsules orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsules.
  Other Names: Zasocitinib
  Arms: TAK-279 Dose 1; TAK-279 Dose 2; TAK-279 Dose 3
Drug: Placebo — TAK-279 placebo-matching capsules.
  Arms: Placebo; TAK-279 Dose 1; TAK-279 Dose 2

SUMMARY:
Crohn's disease (CD) is a long-lasting condition causing inflammation that can affect any part of the gut. The purpose of this study is to evaluate the efficacy and safety of TAK-279 versus placebo in participants with moderately to severely active Crohn's disease (CD). The main aim of this study is to learn if the 3 different doses of TAK-279 reduce bowel inflammation and ulcers in the bowel compared to the placebo after 12 weeks of treatment. Another aim is to compare any medical problems that participants have when they take TAK-279 or placebo and how well the participants tolerate medical problems. An endoscopy will be used to check the bowel for inflammation.

The participants will be treated with TAK-279 for 52 weeks (1 year).

During the study, participants will visit their study clinic 15 times.

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-279. TAK-279 is being tested to treat participants with moderately to severely active Crohn's disease. The study will look at the efficacy and safety of TAK-279.

The study will enroll approximately 268 participants. During the Induction Period participants will be randomly assigned to one of the following treatment groups in a ratio of 1:1:1:1 to receive TAK-279 or placebo which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

1. TAK-279 Dose 1
2. TAK-279 Dose 2
3. TAK-279 Dose 3
4. Placebo

This multi-center trial will be conducted globally. The overall study duration is approximately 60 weeks including a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years old with diagnosis of CD for at least 30 days. In South Korea, the age requirement for adult participants is >=19 years of age.
2. Confirmed diagnosis of moderately to severely active CD assessed by SES-CD and CDAI.
3. Participants must have had an inadequate response to, loss of response to, or intolerance to at least one or more conventional, biologic, or advanced therapy for CD.

Exclusion Criteria:

1. Participants with indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, and diverticular disease associated with colitis, and/or ulcerative colitis.
2. Have complications of CD that might require surgery during the study.
3. Participants with a current ostomy.
4. Participants who have failed 3 or more classes of advanced therapies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2027-07-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Endoscopic Response Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12 | Week 12
  Endoscopic response is defined by decrease in SES-CD >50% from baseline (or for participants with isolated ileal disease, SES-CD <=4 or at least a 2-point reduction from baseline). SES-CD evaluates 4 endoscopic variables (the intestinal surface affected by ulcers, the intestinal surface affected by other inflammatory lesions, the presence of ulcers, and the presence of narrowing).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) at Week 12 | Week 12
  Clinical remission is defined as a CDAI score of <150 points.
Percentage of Participants With a Clinical Response Based on the CDAI at Week 12 | Week 12
  Clinical response is defined as >=100-point decrease from Baseline in CDAI score.
Percentage of Participants Achieving Endoscopic Remission Based on SES-CD at Week 12. | Week 12
  Endoscopic remission as per SES-CD is defined as SES-CD score <=4 or <=2 for ileal disease, no subscore >1.
Percentage of Participants Achieving Clinical Remission in 2-item Patient-reported Outcome Measure (PRO2) at Week 12 | Week 12
  Clinical remission based on PRO2 is defined as average daily liquid or very soft stool frequency (SF) score <=2.8 and not worse than baseline and average daily abdominal pain (AP) score <=1 and not worse than baseline.
Percentage of Participants With a Clinical Response in PRO2 at Week 12 | Week 12
  Clinical response based on PRO2 is defined as >=30% decrease in average daily very soft or liquid stools and/ or >=30% decrease in average AP from baseline.
Percentage of Participants With no Bowel Urgency at Week 12 | Week 12
  Bowel urgency is assessed using a 1-item daily patient diary that asks participants to indicate if they had an urgent bowel movement (when they felt the need to rush to the toilet to avoid an accident) in the past 24 hours. Response options, "Yes" or "No" will be coded as numeric values.
Percentage of Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score >=170 at Week 12 | Week 12
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question will be assessed on a 7-point Likert scale. Each domain score is the sum of 8 responses each ranging from 1 to 7, where 1 indicates worst function and 7 the best. The total score ranges from 32 to 224, with higher scores representing better quality of life.
Change from Baseline in Health-related Quality of Life (HRQoL) as per IBDQ Total Score at Week 12 | Baseline to Week 12
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. Within dimensions, each question will be assessed on a 7-point Likert scale. Each domain score is the sum of 8 responses each ranging from 1 to 7, where 1 indicates worst function and 7 the best. The total score ranges from 32 to 224, with higher scores representing better quality of life.
Change from Baseline in Fatigue as per Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 12 | Baseline to Week 12
  FACIT-Fatigue questionnaire contains 13 fatigue-related questions. The responses to the 13 items on the FACIT-Fatigue questionnaire are each measured on a 5-point Likert scale, where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit and 4=Very much. The total score ranges from 0 to 52. High scores represent less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (176):
- United States (26):
  - GastroIntestinal BioSciences, Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - UCI Health, Orange, California
  - West Central Gastroenterology, LLP, d/b/a/ Gastro Florida, Clearwater, Florida
  - Auzmer Research, Lakeland, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - GI PROS, Inc., Naples, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Emory University Hospital, The Emory Clinic, Atlanta, Georgia
  - Atlanta Center For Gastroenterology, P.C., Decatur, Georgia
  - The University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University Of Louisville, Louisville, Kentucky
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - BVL Clinical Research, Liberty, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - University Gastroenterology Providence, Providence, Rhode Island
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Novel Research, LLC, Bellaire, Texas
  - Texas Digestive Disease Consultants, PLLC d/b/a GI Alliance, Fort Worth, Texas
  - TDDC dba Alliance Research, Mansfield, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Washington Medical Center, Seattle, Washington
- Australia (9):
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Mater Cancer Care Centre-Mater Health Services, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Western Health/Footscray Hospital, Melbourne, Victoria
  - Harry Perkins Medical Research Institute Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Northern Hospital Epping, Epping
  - Sir Charles Gairdner Hospital (SCGH) - Comprehensive Cancer Centre, Nedlands
- Belgium (4):
  - Hopital Universitaire de Bruxelles/ Academisch Ziekenhuis Brussel, Brussels, Anderlecht / Region Capitale de Bruxelles/ Brussel
  - CHU Saint-Pierre - Porte de Hal, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman, Liège
- Bulgaria (6):
  - UMBAL Kaspela, Plovdiv
  - Multi-Profile Hospital for Active Treatment (MHAT) Hadji Dimitar, Sliven
  - Acibadem City clinic Tokuda hospital, Sofia
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia
  - University Hospital Tsaritsa Yoanna - Isul (University Hospital Queen Giovanna), Sofia
  - Acibadem City Clinic Mladost Hospital, Sofia
- Canada (8):
  - Heritage Medical Research Clinic - University Of Calgary, Calgary, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Nova Scotia Health Authority - Queen Elizabeth II Heath Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - University of Toronto - Mount Sinai Hospital - The Lunenfeld-Tanenbaum Research Institute, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Center, Montreal, Quebec
- China (10):
  - Chongqing General Hospital, Chongqing, Chongqing Sheng
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University (SYSU) - The First Affiliated Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - China Medical University (CMU) - Shengjing Hospital (The Second Affiliated Hospital) - Huaxiang Campus, Shenyang, Liaoning
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sun Yat-sen University - The Sixth Affiliated Hospital (Guangdong Gastrointestinal Hospital), Guangzhou
  - Zhejiang University School of Medicine - Sir Run Run Shaw Hospital (SRRSH), Hangzhou
  - Shanghai Pudong New District Zhoupu Hospital, Shanghai
- Czechia (12):
  - NH Hospital, Hořovice, Central Bohemia
  - SurGal Clinic SRO, Brno
  - Vojenska Nemocnice Brno, Brno
  - University Hospital Brno, Brno
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - EndoArt, Ostrava
  - Fakultni Nemocnice Ostrava (FNO), Ostrava-Poruba
  - Gastromedic s.r.o, Pardubice
  - Endohope Clinic, Prague
  - Axon Clinical s.r.o., Prague
  - Masaryk Hospital, Ústí nad Labem
- Denmark (6):
  - Odense Universitetshospital (OUH) (Odense University Hospital), Odense, Region Syddanmark
  - Aalborg Hospital, Aalborg
  - Sydvestjysk Region/Esbjerg Hospital, Esbjerg
  - Hillerod Hospital, Hilleroed Sygehus, Hillerød
  - Hvidovre Hospital Medicinsk Gastroenterologisk Afdeling, Hvidovre
  - Region Sjaelland Sygehus Nord, Koge Sygehus, Køge
- France (5):
  - Centre Hospital Regional Et Universitaire De Tours (Chru Tours) - Houpital Trousseau, Chambray-lès-Tours
  - CHU De Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - Hopital l'Archet 2, Nice
  - Hopital Nord Chu Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Regional Universitaire de Nancy, Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Universitaetsklinik Frankfurt, Frankfurt
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitaetsklinikum Schleswig-Holstein, UKSH-Campus Kiel, Kiel
  - St. Marien- und St. Annastiftskrankenhaus, Ludwigshafen
  - Universitaetsklinikum Mannheim GmbH, Mannheim
  - Universitaetsklinikum Tuebingen, Tübingen
  - University Hospital Of Ulm, Universitatsklinikum Ulm, Ulm
- Greece (6):
  - University General Hospital of Patras, Pátrai, Achaia
  - Evangelismos Hospital, Athens, Attica
  - University of Athens School of Medicine, Alexandra General Hospital, Athens, Attica
  - University Hospital of Heraklion, Heraklion, Crete
  - Sotiria General Hospital of Athens, Athens
  - G.N.A. Gennimatas, Athens
- Hungary (4):
  - Clinexpert, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Mohacsi Korhaz, Mohács
- Israel (5):
  - Soroka Mc, Beersheba
  - Digestive Disease Institute, Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center - The Edmond and Lily Safra Children's Hospital, Ramat Gan
  - The Chaim Sheba Medical Centre, Tel Aviv
- Italy (7):
  - IRCCS - AOU di Bologna - SantOrsola Malpighi, Bologna
  - Fondazione IRCCS Ospedale Maggiore Policlinico Mangiagalli e Regina Elena - Clinica Mangiagalli, Milan
  - Ospedale San Raffaele (HSR) Instituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - A. Gemelli University Hospital, Catholic University of the Sacred Heart, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - IRCCS Istituto clinico humanitas - Humanitas Mirasole spa, Rozzano
- Japan (13):
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - The Jikei University Hospital, Minato, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tsujinaka Hospital Kashiwanoha, Chiba
  - Fukuoka University Hospital, Fukuoka
  - Institute of Science Tokyo Hospital, Tokyo
  - Toyama University Hospital, Toyama
- Netherlands (3):
  - Zuyderland Medisch Centrum - Sittard-Geleen, Geleen, Limburg
  - Amsterdam University Medical Center (Amsterdam UMC), Vrije University Medical Center (VUMC), Amsterdam
  - St. Elisabeth Ziekenhuis, Tilburg
- Norway (2):
  - Akershus University Hospital, Lorenskog, Akershus
  - Oslo Univeristy Hospital Ulleval Hospital, Oslo
- Poland (16):
  - Gastromed Kopon, Zmudzinski i Wspolnicy Sp.j. Specjalistyczne Centrum Gastrologii i Endoskopii Specjalistyczne Gabinety Lekarskie, Torun, Kujawsko-pomo
  - Centrum Medyczne Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - PlanetMed Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA, Warsaw, Masovian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Manermed Sp. z o.o - CM Medis, Bydgoszcz
  - Oddzial Kliniczny Gastroenterologii Ogolnej i Onkologicznej SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Centrum Medyczne Med-Gastr, Lodz
  - Medrise sp. z o.o, Lublin
  - Centrum Medyczne Medyk Sp. z o.o. Sp. K., Rzeszów
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - H-T. Centrum Medyczne Sp. z o.o. Sp.k., Tychy
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
  - ETG Zamosc, Zamość
  - AmiCare Sp. z o.o. Sp. k., Lodz, Łódź Voivodeship
- Romania (6):
  - Policlinica Algomed: Centrul De Gastroenterologie Dr. Goldis, Timișoara, Jud Timis
  - Clinical Hospital Colentina-Spitalul Clinic Colentina, Bucharest
  - Clinica Medicum, Bucharest
  - Spital Clinic Dr I Cantacuzino, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Euroclinic, Bucharest
- Slovakia (5):
  - Fakultna nemocnica F. D. Roosevelta, Banská Bystrica
  - Cliniq s. r. o., Bratislava
  - Endomed, Košice
  - Fakultna Nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Accout Center, s.r.o.- Gastroenterologicka ambulancia, Šahy
- South Korea (7):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center (AMC), Seoul
  - Samsung Medical Center, Seoul
- Switzerland (2):
  - University Hospital Basel, Basel
  - Intesto - Gastroenterologische Praxis & Crohn-Colitis-Zentrum Bern, Bern
- Taiwan (3):
  - Changhua Christian Hospital, Changhua, Changhua County
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - China Medical University Hospital, Taichung
- United Kingdom (4):
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Wingate Institute for Neurogastroenterology, Wingate Clinical Trials Facility, Barts Health NHS Trust, London, E1 2at
  - South Eastern Health and Social Care Trust - The Ulster Hospital, Belfast
  - St Thomas' Hospital - Guy's & St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/6b7fad105d7b4f53?idFilter=%5B%22TAK-279-CD-2001%22%5D